CLINICAL TRIAL: NCT01696136
Title: Multi-electrode PulmonarY Vein Isolation Versus Single Tip Wide Area Catheter Ablation for PAF a Randomized Multinational Multicenter Trial
Brief Title: Multi-electrode PulmonarY Vein Isolation Versus Single Tip Wide Area Catheter Ablation for Paroxysmal Atrial Fibrillation (PAF)
Acronym: MYSTIC-PAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: L.V.A. Boersma (Other)
Responsible Party: Sponsor-Investigator, L.V.A. Boersma, Cardiologist, R&D Cardiologie
Organization: R&D Cardiologie (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RDC-2010.01
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Atrial Fibrillation
Keywords: Ablation; Multi-electrode catheter; Single-tip catheter; Holter
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AF-Ablation with Multi-electrode catheter (Active Comparator): Regular AF-ablation with a multi-electrode ablation catheter
  Interventions: Device: Cardiac ablation for Atrial Fibrillation
- AF-Ablation with single-tip electrode (Active Comparator): Regular AF-ablation with a regular single-tip ablation catheter
  Interventions: Device: Cardiac ablation for Atrial Fibrillation

INTERVENTIONS:
Device: Cardiac ablation for Atrial Fibrillation — Cardiac ablation for Atrial Fibrillation

SUMMARY:
The MYSTIC_PAF trial investigates the differences between treatment with a single-tip catheter against a multielectrode catheter in cardiac ablation procedures in patients with paroxysmal atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. History of symptomatic paroxysmal atrial fibrillation defined as:

   * Self-terminating AF with episodes lasting no more than seven consecutive days before spontaneous conversion back to sinus rhythm
   * Documentation of one or more events with PAF tracings by ECG, event recordings, pacemaker strips or monitor rhythm strips within the past year
   * AF symptoms defined as the manifestation of any of the following:

     * Palpitations
     * Fatigue
     * Exertional dyspnea
     * Effort intolerance
2. Age between 18 and 70
3. Willingness, ability and commitment to participate in baseline and follow-up evaluations for the full length of the study

Exclusion Criteria:

1. Structural heart disease of clinical significance including:

   * Previous cardiac surgery (excluding CABG)
   * Symptoms of congestive heart failure including, but not limited to, NYHA Class III or IV CHF and/or documented ejection fraction < 40% measured by acceptable cardiac testing
   * Left atrial diameter of > 50mm as measured in the parasternal long axis on transthoracic echocardiogram
   * Stable/unstable angina or ongoing myocardial ischemia
   * Myocardial infarction (MI) within three months of enrollment
   * Aortic or mitral valve disease > Grade II
   * Congenital heart disease (not including ASD or PFO without a right to left shunt) where the underlying abnormality increases the risk of an ablative procedure
   * Prior ASD or PFO closure with a device using a percutaneous approach
   * Hypertrophic cardiomyopathy (LV wall thickness > 1.5 cm)
   * Pulmonary hypertension (mean or systolic PA pressure >50mm Hg on Doppler echo
2. Prior ablation for arrhythmias other than AF within the past three months
3. Prior left sided AF ablation
4. Enrollment in any other ongoing arrhythmia study protocol Any ventricular tachyarrhythmias currently being treated where the arrhythmia or the management may interfere with this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Freedom of AF | Month 3 after intervention
  Is the patient free of Atrial Fibrillation, at month 3 after the ablation intervention, and not taking anti-arrhythmic drugs

CONTACTS AND LOCATIONS:
Locations (1):
- St. Antonius Ziekenhuis Nieuwegein, Nieuwegein, Utrecht, Netherlands

REFERENCES:
- [Derived] Boersma LV, van der Voort P, Debruyne P, Dekker L, Simmers T, Rossenbacker T, Balt J, Wijffels M, Degreef Y. Multielectrode Pulmonary Vein Isolation Versus Single Tip Wide Area Catheter Ablation for Paroxysmal Atrial Fibrillation: A Multinational Multicenter Randomized Clinical Trial. Circ Arrhythm Electrophysiol. 2016 Apr;9(4):e003151. doi: 10.1161/CIRCEP.115.003151. PMID 27071830